CLINICAL TRIAL: NCT02874794
Title: A Multicenter, Randomized, Double-blind, Double-dummy, Parallel Group, Active-controlled, Forced-titration, 12-week Comparison of Combined Angiotensin-neprilysin Inhibition With Sacubitril and Valsartan Versus Enalapril on Changes in Central Aortic Stiffness in Patients With Heart Failure and Reduced Ejection Fraction (HFrEF)
Brief Title: Study of Effects of Sacubitril/Valsartan vs. Enalapril on Aortic Stiffness in Patients With Mild to Moderate HF With Reduced Ejection Fraction
Acronym: EVALUATE-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLCZ696BUS08
Record Dates: First submitted 2016-08-05; First posted 2016-08-22 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure and Reduced Ejection Fraction
Keywords: Heart Failure; Reduced Ejection Fraction; Central Aortic Stiffness; Vascular; Echocardiogram; Aortic Stiffness
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; sacubitril; Valsartan; Enalapril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCZ696 (sacubitril/valsartan) (Experimental): minimum dose: 24/26mg, BID, oral, tablet maximum dose: 97/103mg, BID, oral, tablet All patients will begin on Dose Level 1 (24/26mg) and will be titrated every two weeks to target Dose level 3 (97/103mg). LCZ696 tablets will be provided for the 12-week open label extension.
  Interventions: Drug: LCZ696 (sacubitril/valsartan); Drug: Placebo of Enalapril
- Enalapril (Active Comparator): minimum dose: 2.5mg, BID, oral, tablet maximum dose: 10 mg, BID, oral tablet All patients will begin on Dose Level 1 (2.5mg) and will be titrated every two weeks to target Dose level 3 (10mg).
  Interventions: Drug: Enalapril; Drug: Placebo of LCZ696

INTERVENTIONS:
Drug: LCZ696 (sacubitril/valsartan) — 24/26mg, 49/51mg and 97/103mg oral, tablets.
  Other Names: LCZ696
  Arms: LCZ696 (sacubitril/valsartan)
Drug: Enalapril — 2.5mg, 5mg, and 10mg, oral, tablets
  Arms: Enalapril
Drug: Placebo of Enalapril — matching placebo (2.5mg, 5mg and 10mg) oral, tablets
  Arms: LCZ696 (sacubitril/valsartan)
Drug: Placebo of LCZ696 — matching placebo (24/26mg, 49/51mg and 97/103mg) oral, tablets
  Arms: Enalapril

SUMMARY:
To determine whether treatment with sacubitril/valsartan provides a superior effect on aortic characteristic impedance compared to enalapril in patients with heart failure and reduced ejection fraction (left ventricular ejection fraction [LVEF] ≤ 40%) after 12 weeks of treatment. The primary endpoint is the change in aortic characteristic impedance (Zc = dP/dQ in early systole) between baseline and Week 12.

ELIGIBILITY:
Inclusion Criteria:

* History of HTN and one of the following at BOTH screening and pre-randomization:

  1. SBP >105 mm Hg on antihypertensive medication.
  2. SBP >/= 140 mm Hg and NOT on antihypertensive medication.
* NYHA class I-III heart failure and with reduced ejection fraction </= 40%, as determined by any local measurement made within the past 12 months using echocardiography, MUGA, CT scanning, MRI, ventricular angiography or single-photon emission computed tomography (SPECT), provided no subsequent measurement above 40%. Patients who have had an intervening medical event (e.g. myocardial infarction) or procedure (e.g. revascularization, cardiac resynchronization), must have a reassessment of EF ≥ 3 months following the event to ensure that eligibility criteria are still met.
* On stable doses of treatment with guideline-directed therapy, other than ACEis and ARBs prior to randomization.

  1. If the patient is currently taking an ACEi, a 36-hour washout is required prior to randomization (Visit 2).
  2. If the patient is currently taking an ARB, they must discontinue the ARB before initiation of study treatment however washout is not required.
* On an optimal medical regiment of diuretics and background medications to effectively treat co-morbidities such as HTN, DM, and coronary artery disease.

Key Exclusion Criteria:

* History of hypersensitivity to any of the study drigs, including history of hypersensitivity to drugs of similar chemical classes, or allergy to ACEis, ARBs, or NEP inhibitors as well as known or suspected contraindications to the study drugs.
* Previous history of intolerance to sacubitril and valsartan, ACEi or ARB standard of care doses despite appropriate and gradual up-titration.
* History of angioedema, drug-related or otherwise.
* Requirement of treatment with both ACE inhibitor and ARB.
* Current or prior treatment with sacubitril and valsartan.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2019-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (72):
- United States (72):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Newport Beach, California
  - Novartis Investigative Site, Northridge, California
  - Novartis Investigative Site, Santa Ana, California
  - Novartis Investigative Site, Van Nuys, California
  - Novartis Investigative Site, Greenwich, Connecticut
  - Novartis Investigative Site, Norwalk, Connecticut
  - Novartis Investigative Site, Stamford, Connecticut
  - Novartis Investigative Site, Trumbull, Connecticut
  - Novartis Investigative Site, Newark, Delaware
  - Novartis Investigative Site, Atlantis, Florida
  - Novartis Investigative Site, Aventura, Florida
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Coral Gables, Florida
  - Novartis Investigative Site, Daytona Beach, Florida
  - Novartis Investigative Site, Doral, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Hialeah, Florida
  - Novartis Investigative Site, Inverness, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Jupiter, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Naples, Florida
  - Novartis Investigative Site, Saint Augustine, Florida
  - Novartis Investigative Site, Athens, Georgia
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Blue Ridge, Georgia
  - Novartis Investigative Site, Eatonton, Georgia
  - Novartis Investigative Site, Macon, Georgia
  - Novartis Investigative Site, Coeur d'Alene, Idaho
  - Novartis Investigative Site, Fairview Heights, Illinois
  - Novartis Investigative Site, Gurnee, Illinois
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Eunice, Louisiana
  - Novartis Investigative Site, Minden, Louisiana
  - Novartis Investigative Site, Monroe, Louisiana
  - Novartis Investigative Site, Slidell, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Alpena, Michigan
  - Novartis Investigative Site, Owosso, Michigan
  - Novartis Investigative Site, Saginaw, Michigan
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Hillsborough, New Jersey
  - Novartis Investigative Site, Linden, New Jersey
  - Novartis Investigative Site, Manalapan, New Jersey
  - Novartis Investigative Site, Mountain Lakes, New Jersey
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, Lake Success, New York
  - Novartis Investigative Site, Rosedale, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Greenville, North Carolina
  - Novartis Investigative Site, Lenoir, North Carolina
  - Novartis Investigative Site, Yardley, Pennsylvania
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Amarillo, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, McKinney, Texas
  - Novartis Investigative Site, Sherman, Texas
  - Novartis Investigative Site, Tomball, Texas
  - Novartis Investigative Site, Webster, Texas
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Richland, Washington
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, Manitowoc, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Lee S, Claggett BL, Fang JC, Mitchell GF, Ward JH, Solomon SD, Skali H, Desai AS, Hegde SM. Changes in cardiac structure and function are associated with health-related quality of life in heart failure patients with reduced ejection fraction: Results from the EVALUATE-HF trial. Eur J Heart Fail. 2025 Nov;27(11):2582-2593. doi: 10.1002/ejhf.3760. Epub 2025 Jul 18. PMID 40678912
- [Derived] Myhre PL, Claggett BL, Shah AM, Prescott MF, Ward JH, Fang JC, Mitchell GF, Solomon SD, Desai AS. Changes in cardiac biomarkers in association with alterations in cardiac structure and function, and health status in heart failure with reduced ejection fraction: the EVALUATE-HF trial. Eur J Heart Fail. 2022 Jul;24(7):1200-1208. doi: 10.1002/ejhf.2541. Epub 2022 May 30. PMID 35560696
- [Derived] Myhre PL, Prescott MF, Murphy SP, Fang JC, Mitchell GF, Ward JH, Claggett B, Desai AS, Solomon SD, Januzzi JL. Early B-Type Natriuretic Peptide Change in HFrEF Patients Treated With Sacubitril/Valsartan: A Pooled Analysis of EVALUATE-HF and PROVE-HF. JACC Heart Fail. 2022 Feb;10(2):119-128. doi: 10.1016/j.jchf.2021.09.007. Epub 2022 Jan 12. PMID 35115085
- [Derived] Mitchell GF, Solomon SD, Shah AM, Claggett BL, Fang JC, Izzo J, Abbas CA, Desai AS; EVALUATE-HF Investigators*. Hemodynamic Effects of Sacubitril-Valsartan Versus Enalapril in Patients With Heart Failure in the EVALUATE-HF Study: Effect Modification by Left Ventricular Ejection Fraction and Sex. Circ Heart Fail. 2021 Mar;14(3):e007891. doi: 10.1161/CIRCHEARTFAILURE.120.007891. Epub 2021 Mar 5. PMID 33663237
- [Derived] Desai AS, Solomon SD, Shah AM, Claggett BL, Fang JC, Izzo J, McCague K, Abbas CA, Rocha R, Mitchell GF; EVALUATE-HF Investigators. Effect of Sacubitril-Valsartan vs Enalapril on Aortic Stiffness in Patients With Heart Failure and Reduced Ejection Fraction: A Randomized Clinical Trial. JAMA. 2019 Sep 17;322(11):1077-1084. doi: 10.1001/jama.2019.12843. PMID 31475296
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=514

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 892 patients screened for the study, 465 completed screening and were enrolled. Of the 465 randomized, 1 patient was randomized in error to the sacubitril/valsartan group and was not treated. The Full Analysis Set and Safety Set are based on 464 patients who received treatment.
Groups:
- Enalapril (Double-Blind Phase): minimum dose: 2.5mg, BID, oral, tablet. maximum dose: 10 mg, BID, oral tablet. All patients began on Dose Level 1 (2.5mg) and were titrated every two weeks to target Dose level 3 (10mg).
- Sacubitril/Valsartan (Double-Blind Phase): minimum dose: 24/26mg, BID, oral, tablet. maximum dose: 97/103mg, BID, oral, tablet. All patients began on Dose Level 1 (24/26mg) and were titrated every two weeks to target Dose level 3 (97/103mg).
Period: Overall Study
Arm/Group | Enalapril (Double-Blind Phase) | Sacubitril/Valsartan (Double-Blind Phase)
Started | 233 | 232
Completed | 226 | 221
Not Completed | 7 | 11
Not completed — Physician Decision | 3 | 2
Not completed — Withdrawal by Subject | 2 | 8
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Enalapril (Double-Blind Phase) | Sacubitril/Valsartan (Double-Blind Phase) | Total
Number analyzed (Participants) | 233 | 231 | 464
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 90 | 190
  >=65 years | 133 | 141 | 274
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 61 | 109
  Male | 185 | 170 | 355
Race/Ethnicity, Customized [Number; unit: articipants]
  Caucasian (White) | 175 | 166 | 341
  Black | 53 | 62 | 115
  Asian | 2 | 2 | 4
  Native American | 1 | 0 | 1
  Other | 0 | 1 | 1
  Unknown | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Aortic Characteristic Impedance at Week 12
Description: Aortic characteristic impedance, Zc, is the ratio of the change in pressure (dP)produced by a given change in flow (dQ) in early systole, i.e., Zc = dP/dQ. Zc is related directly to aortic wall stiffness and inversely to lumen area.
Time Frame: Baseline, Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: dyne x sec/cm5
Arm/Group | Enalapril (Double-Blind Phase) | Sacubitril/Valsartan (Double-Blind Phase)
Number analyzed (Participants) | 233 | 231
dyne x sec/cm5 | -0.7 (5.5) | -2.9 (5.5)
Statistical Analysis 1: Comparison: Enalapril (Double-Blind Phase) vs Sacubitril/Valsartan (Double-Blind Phase); Test type: Superiority; p = 0.7827, ANCOVA; Median Difference (Final Values) = -2.2, 95% CI 2-sided [-17.6 to 13.2]

2. Secondary Outcome: Pearson Correlation Coefficient Between Change From Baseline in Aortic Characteristic Impedance and Biomarker Levels: B-type Natriuretic Peptide (BNP) During Both Trough and 4 Hours Post-dose at Week 4
Description: Pearson correlation coefficients between changes from baseline in aortic characteristic impedance (dyne x sec/cm5) and biomarker levels such as BNP (pg/ML) during both trough and 4 hours post-dose at Week 4
Time Frame: Pre-dose and 4 hours post dose at week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Pearson's Correlation
Arm/Group | Enalapril (Double-Blind Phase) | Sacubitril/Valsartan (Double-Blind Phase)
Number analyzed (Participants) | 233 | 231
Pearson's Correlation
  Week 4 (pre-dose): number analyzed (Participants) | 213 | 200
  Week 4 (pre-dose) | 0.022 [-0.113 to 0.156] | 0.070 [-0.069 to 0.207]
  Week 4 (post-dose): number analyzed (Participants) | 193 | 188
  Week 4 (post-dose) | -0.127 [-0.263 to 0.015] | 0.016 [-0.128 to 0.159]

3. Secondary Outcome: Pearson Correlation Coefficient Between Change From Baseline in Aortic Characteristic Impedance and Biomarker Levels: cGMP/U-creatinine During Both Trough and 4 Hours Post-dose at Week 4
Description: Pearson correlation coefficient between changes from baseline in aortic characteristic impedance (dyne x sec/cm5) and biomarker levels such as U-cGMP/U-creatinine ratio (nmol/mmol) during both trough and 4 hours post-dose at Week 4
Time Frame: pre-dose and 4 hours post dose at week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Pearson's correlation coefficient
Arm/Group | Enalapril (Double-Blind Phase) | Sacubitril/Valsartan (Double-Blind Phase)
Number analyzed (Participants) | 233 | 231
Pearson's correlation coefficient
  Week 4 (pre-dose): number analyzed (Participants) | 209 | 196
  Week 4 (pre-dose) | 0.087 [-0.049 to 0.220] | 0.098 [-0.043 to 0.235]
  Week 4 (post-dose): number analyzed (Participants) | 193 | 186
  Week 4 (post-dose) | 0.110 [-0.032 to 0.247] | 0.157 [0.014 to 0.294]

4. Secondary Outcome: Change From Baseline in N-terminal Pro-brain Natriuretic Peptide (NT-proBNP)
Description: Change from baseline in N-terminal pro-brain natriuretic peptide (NT-proBNP)
Time Frame: Baseline, Week 12
Population: Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Enalapril (Double-Blind Phase) | Sacubitril/Valsartan (Double-Blind Phase)
Number analyzed (Participants) | 233 | 231
pg/mL | 0.9500 [0.8673 to 1.0406] | 0.6334 [0.5778 to 0.6944]
Statistical Analysis 1: Comparison: Enalapril (Double-Blind Phase) vs Sacubitril/Valsartan (Double-Blind Phase); Test type: Superiority; p < .0001, ANCOVA; Ratio of Geometric Means = 0.6667, 95% CI 2-sided [0.5858 to 0.7589]

5. Secondary Outcome: Change From Baseline in Echocardiographic Measure: Global Longitudinal Strain
Description: Parameter measured by echocardiography.
Time Frame: Baseline, Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Enalapril (Double-Blind Phase) | Sacubitril/Valsartan (Double-Blind Phase)
Number analyzed (Participants) | 233 | 231
Percentage | -0.21 (0.16) | -0.34 (0.16)
Statistical Analysis 1: Comparison: Enalapril (Double-Blind Phase) vs Sacubitril/Valsartan (Double-Blind Phase); Test type: Superiority; p = 0.5792, ANCOVA; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.58 to 0.33]

6. Secondary Outcome: Change From Baseline in Echocardiographic Measure: Left Atrial Volume Index (LAVi)
Description: Parameter measured by echocardiography
Time Frame: Baseline, Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mL/m2
Arm/Group | Enalapril (Double-Blind Phase) | Sacubitril/Valsartan (Double-Blind Phase)
Number analyzed (Participants) | 233 | 231
mL/m2 | 0.63 (0.44) | -2.17 (0.44)
Statistical Analysis 1: Comparison: Enalapril (Double-Blind Phase) vs Sacubitril/Valsartan (Double-Blind Phase); Test type: Superiority; p < .0001, ANCOVA; Mean Difference (Final Values) = -2.80, 95% CI 2-sided [-4.02 to -1.59]

7. Secondary Outcome: Change From Baseline in Echocardiographic Measure: Mitral Annular E' Velocity (Doppler Tissue Imaging)
Description: Parameter measured by echocardiography
Time Frame: Baseline, Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: cm/sec
Arm/Group | Enalapril (Double-Blind Phase) | Sacubitril/Valsartan (Double-Blind Phase)
Number analyzed (Participants) | 233 | 231
cm/sec | -0.00 (0.11) | -0.03 (0.11)
Statistical Analysis 1: Comparison: Enalapril (Double-Blind Phase) vs Sacubitril/Valsartan (Double-Blind Phase); Test type: Superiority; p = 0.8617, ANCOVA; Median Difference (Final Values) = -0.03, 95% CI 2-sided [-0.33 to 0.27]

8. Secondary Outcome: Change From Basekine in Echocardiographic Measure: Mitral E/E'
Description: Parameter measured by echocardiography
Time Frame: Baseline, Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Enalapril (Double-Blind Phase) | Sacubitril/Valsartan (Double-Blind Phase)
Number analyzed (Participants) | 233 | 231
Ratio | 0.32 (0.36) | -1.43 (0.36)
Statistical Analysis 1: Comparison: Enalapril (Double-Blind Phase) vs Sacubitril/Valsartan (Double-Blind Phase); vs Enalapril; Test type: Superiority; p = 0.0007, ANCOVA; Median Difference (Final Values) = -1.75, 95% CI 2-sided [-2.76 to -0.75]

9. Secondary Outcome: Change From Baseline in Echocardiographic Measure: Left Ventricular Ejection Fraction (LVEF)
Description: Parameter measured by echocardiography
Time Frame: Baseline, Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Sacubitril/Valsartan (Double-Blind Phase) | Enalapril (Double-Blind Phase)
Number analyzed (Participants) | 233 | 231
Percentage | 1.30 (0.37) | 1.94 (0.38)
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (Double-Blind Phase) vs Enalapril (Double-Blind Phase); Test type: Superiority; p = 0.2354, ANCOVA; Median Difference (Final Values) = 0.63, 95% CI 2-sided [-0.41 to 1.68]

10. Secondary Outcome: Change From Baseline in Echocardiographic Measure: Ventricular-vascular Coupling (Ea/Ees)
Description: Parameter measured by echocardiography
Time Frame: Baseline, Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Ea/Ees Ratio
Arm/Group | Enalapril (Double-Blind Phase) | Sacubitril/Valsartan (Double-Blind Phase)
Number analyzed (Participants) | 233 | 231
Ea/Ees Ratio | 0.03 (0.01) | 0.02 (0.02)
Statistical Analysis 1: Comparison: Enalapril (Double-Blind Phase) vs Sacubitril/Valsartan (Double-Blind Phase); Test type: Superiority; p = 0.8215, ANCOVA; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.05 to 0.04]

11. Secondary Outcome: Change From Baseline in Echocardiographic Measure: Left Ventricular End Systolic Volume Index (LVESVi)
Description: Parameter measured by echocardiography
Time Frame: Baseline, Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mL/m2
Arm/Group | Enalapril (Double-Blind Phase) | Sacubitril/Valsartan (Double-Blind Phase)
Number analyzed (Participants) | 233 | 231
mL/m2 | -3.28 (0.55) | -4.86 (0.56)
Statistical Analysis 1: Comparison: Enalapril (Double-Blind Phase) vs Sacubitril/Valsartan (Double-Blind Phase); Test type: Superiority; p = 0.0452, ANCOVA; Median Difference (Final Values) = -1.58, 95% CI 2-sided [-3.13 to -0.03]

12. Secondary Outcome: Change From Baseline in Echocardiographic Measure: Left Ventricular End Diastolic Volume Index (LVEDVi)
Description: Parameter measured by echocardiography
Time Frame: Baseline, Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mL/m2
Arm/Group | Enalapril (Double-Blind Phase) | Sacubitril/Valsartan (Double-Blind Phase)
Number analyzed (Participants) | 233 | 231
mL/m2 | -3.18 (0.61) | -5.15 (0.62)
Statistical Analysis 1: Comparison: Enalapril (Double-Blind Phase) vs Sacubitril/Valsartan (Double-Blind Phase); Test type: Superiority; p = 0.0242, ANCOVA; Mean Difference (Final Values) = -1.97, 95% CI 2-sided [-3.68 to -0.26]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment, plus 30 days post treatment, up to maximum duration of approximately 2.5 years.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Groups:
- Double Blind Phase Enalapril: Minimum dose: 2.5mg, BID, oral, tablet. Maximum dose: 10 mg, BID, oral tablet. All patients began on Dose Level 1 (2.5mg) and were titrated every two weeks to target Dose level 3 (10mg).
- Double Blind Phase Sacubitril/Valsartan: Minimum dose: 24/26mg, BID, oral, tablet. Maximum dose:
  97/103mg, BID, oral, tablet. All patients began on Dose Level 1 (24/26mg) and were titrated every two weeks to target Dose level 3 (97/103mg).
- Open-Label Phase Sacubitril/Valsartan: LCZ696 tablets were provided for the 12-week open label extension.
Arm/Group | Double Blind Phase Enalapril | Double Blind Phase Sacubitril/Valsartan | Open-Label Phase Sacubitril/Valsartan
All-Cause Mortality (participants affected / at risk) | 1/233 | 1/231 | 5/454
Serious Adverse Events (participants affected / at risk) | 21/233 | 17/231 | 40/454
Other Adverse Events (participants affected / at risk) | 32/233 | 43/231 | 42/454
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind Phase Enalapril (N=233) | Double Blind Phase Sacubitril/Valsartan (N=231) | Open-Label Phase Sacubitril/Valsartan (N=454)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 3
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 0 | 2
Cardiac failure (Cardiac disorders) | 3 | 1 | 2
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 3
Cardiac failure congestive (Cardiac disorders) | 2 | 1 | 3
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 2 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Necrosis (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Swelling (General disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1 | 2
Sepsis (Infections and infestations) | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carotid artery disease (Nervous system disorders) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 1
Device failure (Product Issues) | 0 | 0 | 1
Device malfunction (Product Issues) | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Dry gangrene (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind Phase Enalapril (N=233) | Double Blind Phase Sacubitril/Valsartan (N=231) | Open-Label Phase Sacubitril/Valsartan (N=454)
Hyperkalaemia (Metabolism and nutrition disorders) | 13 | 17 | 12
Dizziness (Nervous system disorders) | 9 | 13 | 15
Hypotension (Vascular disorders) | 13 | 19 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT02874794/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT02874794/SAP_001.pdf